CLINICAL TRIAL: NCT02686151
Title: The Randomized Clinical Trials of Letrozole Administration During Luteal Phase in Patients Who Have the Risk of Ovarian Hyperstimulation Syndrome
Brief Title: The Letrozole Administration During Luteal Phase
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Bhsu
Record Dates: First submitted 2015-08-20; First posted 2016-02-19 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: Letrozole; OHSS
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Letrozole; Polygeline; Sodium Chloride; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letrozole (Active Comparator): 2.5mg/tablet(Jiangsu Hengrui Medicine Co., Ltd. products), orally taken 5mg once a day for 5 days
  Interventions: Drug: Letrozole
- Polygeline Injection (Other): 500ml and 0.9% Sodium Chloride Injection (250ml) with dexamethasone 1mg intravenous injection，once a day for 2 days
  Interventions: Drug: Polygeline; Drug: Sodium Chloride; Drug: dexamethasone

INTERVENTIONS:
Drug: Letrozole — used after oocyte retrieval
  Other Names: Femara
  Arms: letrozole
Drug: Polygeline — used after oocyte retrieval
  Other Names: polyegline
  Arms: Polygeline Injection
Drug: Sodium Chloride — used after oocyte retrieval
  Other Names: Natrum muriaticum
  Arms: Polygeline Injection
Drug: dexamethasone — used after oocyte retrieval
  Other Names: dexametona
  Arms: Polygeline Injection

SUMMARY:
To investigate the effect of letrozole in patients who have high risk of ovarian hyperstimulation syndrome (OHSS) after oocyte retrieval, the incidence of OHSS were calculated between letrozole group and supporting treatment group.

DETAILED DESCRIPTION:
1. Object:

   Infertility patients who frozen all embryos due to the risk of OHSS were randomized allocated to letrozole or polygeline injection group. Inclusion criteria meet one of the following conditions: (1) oocyte is more than or equal to 20; (2) human chorionic gonadotropin (hCG) injection on serum estradiol levels greater than or equal to 5000 pmol/L; (3) on the day of oocyte unilateral or bilateral ovarian diameter greater than or equal to 10 cm (4) follicle puncture is larger than or equal to number 20. After the informed consent was signed, letrozole or polygeline injection was randomized allocated after oocyte retrieval. OHSS was determined according to Golan diagnosis standards.
2. Clinical data:

   Including age, infertility duration, body mass index (BMI), basic follicle-stimulating hormone (FSH) and luteinizing hormone (LH), antral follicle number (AFC), Gn dosage, estradiol level on hCG injection day, the number of oocytes, the number of embryos, early onset OHSS incidence, and the existence of ascites.
3. Reproductive hormone levels:

1, 4, 7, days after taken letrozole, and the supernatant was collected for serum reproductive hormone test.

ELIGIBILITY:
Inclusion criteria:

1. oocyte is more than or equal to 20;
2. hCG injection on serum estradiol levels greater than or equal to 5000 pmol/L; 3. on the day of oocyte unilateral or bilateral ovarian diameter greater than or equal to 10 cm;

4. follicle puncture is larger than or equal to number 20.

Exclusion criteria:

Allergic to the letrozole or polygeline.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of early OHSS | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, PhD, Principal Investigator — Inner Mongolia Medical University affiliated Hospital; Xiujuan Chen, MD, Principal Investigator — Inner Mongolia Medical University affiliated Hospital
Locations (1):
- The Affiliated Hospital of Inner Mongolia Medical University, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He Q, Xu J, Cui S, Li H, Zhang C. [Relationship between letrozole administration during the luteal phase after oocyte retrieval and the early-stage ovarian hyperstimulation syndrome oocurrence]. Zhonghua Fu Chan Ke Za Zhi. 2014 Dec;49(12):909-13. Chinese. PMID 25608991
- [Background] Wang YQ, Yang J, Xu WM, Xie QZ, Yan WJ, Yin TL, Cheng D, Xiao ZN, Li J. [Luteal letrozole administration decreases serum estrogen level but not the risk of ovarian hyperstimulation syndrome]. Beijing Da Xue Xue Bao Yi Xue Ban. 2013 Dec 18;45(6):869-72. Chinese. PMID 24343064
- [Background] Wiwanitkit V. Letrozole and gonadotropins versus luteal estradiol and GnRH-antagonist protocol: additional concerns. Fertil Steril. 2011 Jun 30;95(8):e78; author reply e80. doi: 10.1016/j.fertnstert.2011.05.009. Epub 2011 May 24. No abstract available. PMID 21605857
- [Background] Elassar A, Engmann L, Nulsen J, Benadiva C. Letrozole and gonadotropins versus luteal estradiol and gonadotropin-releasing hormone antagonist protocol in women with a prior low response to ovarian stimulation. Fertil Steril. 2011 Jun;95(7):2330-4. doi: 10.1016/j.fertnstert.2011.03.103. Epub 2011 Apr 22. PMID 21514582
- [Background] Montville CP, Khabbaz M, Aubuchon M, Williams DB, Thomas MA. Luteal support with intravaginal progesterone increases clinical pregnancy rates in women with polycystic ovary syndrome using letrozole for ovulation induction. Fertil Steril. 2010 Jul;94(2):678-83. doi: 10.1016/j.fertnstert.2009.03.088. Epub 2009 Jun 9. PMID 19515366
- [Background] Fatemi HM, Popovic-Todorovic B, Donoso P, Papanikolaou E, Smitz J, Devroey P. Luteal phase oestradiol suppression by letrozole: a pilot study in oocyte donors. Reprod Biomed Online. 2008 Sep;17(3):307-11. doi: 10.1016/s1472-6483(10)60212-x. PMID 18764999
- [Background] Garcia-Velasco JA, Quea G, Piro M, Mayoral M, Ruiz M, Toribio M, Requena A. Letrozole administration during the luteal phase after ovarian stimulation impacts corpus luteum function: a randomized, placebo-controlled trial. Fertil Steril. 2009 Jul;92(1):222-5. doi: 10.1016/j.fertnstert.2008.04.042. Epub 2008 Aug 16. PMID 18710719
- [Background] Sh Tehrani Nejad E, Abediasl Z, Rashidi BH, Azimi Nekoo E, Shariat M, Amirchaghmaghi E. Comparison of the efficacy of the aromatase inhibitor letrozole and clomiphen citrate gonadotropins in controlled ovarian hyperstimulation: a prospective, simply randomized, clinical trial. J Assist Reprod Genet. 2008 May;25(5):187-90. doi: 10.1007/s10815-008-9209-2. Epub 2008 Apr 19. PMID 18427974
- [Background] Ortiz ME, Ortiz RE, Garfield R, Zepeda AJ, Croxatto HB. Progesterone, but not luteal estrogen, is required for the establishment of pregnancy in the new world monkey Cebus apella. Am J Primatol. 2007 Oct;69(10):1131-40. doi: 10.1002/ajp.20408. PMID 17387700
- [Background] Barroso G, Menocal G, Felix H, Rojas-Ruiz JC, Arslan M, Oehninger S. Comparison of the efficacy of the aromatase inhibitor letrozole and clomiphene citrate as adjuvants to recombinant follicle-stimulating hormone in controlled ovarian hyperstimulation: a prospective, randomized, blinded clinical trial. Fertil Steril. 2006 Nov;86(5):1428-31. doi: 10.1016/j.fertnstert.2006.03.044. Epub 2006 Sep 14. PMID 16978619
- [Background] Fatemi HM, Kolibianakis E, Tournaye H, Camus M, Van Steirteghem AC, Devroey P. Clomiphene citrate versus letrozole for ovarian stimulation: a pilot study. Reprod Biomed Online. 2003 Nov;7(5):543-6. doi: 10.1016/s1472-6483(10)62070-6. PMID 14680546